CLINICAL TRIAL: NCT03383601
Title: A 5-year Cohort Observational Study to Evaluate Frequency of Exacerbations, Respiratory Symptoms, Physical Exercise Intolerance and Abnormal Lung Functions Among Participants Who Use IQOS With Heatsticks Compared to Smokers of Conventional Cigarettes
Brief Title: Сohort Study to Evaluate Exacerbations, Respiratory Symptoms, Physical Exercise Intolerance and Lung Functions Among Participants Who Use IQOS With Heatsticks Compared to Smokers of Conventional Cigarettes
Status: Completed | Type: Observational
Sponsor: Kazakhstan Academy of Preventive Medicine (Other)
Collaborators: Philip Morris International (Industry); Synergy Research Group (Industry); HealthCity LLP (Unknown)
Responsible Party: Sponsor
Other Study IDs: PMI.IIS.2016.1.1.
Record Dates: First submitted 2017-12-07; First posted 2017-12-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Physical Disability; Respiratory Disease
Keywords: COPD; Exacerbation of respiratory symptoms; Functional exercise capacity; Heated Tobacco Products; Respiratory symptoms
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Respiration Disorders; Signs and Symptoms, Respiratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood testing for: complete blood count (CBC), blood cholesterol level, HDL (highdensity lipoprotein), LDL (low-density lipoproteins), triglycerides, C-reactive protein, fibrinogen, glucose. Biomarker testing for sRAGE, ICAM1, CCL20 and probably other biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Users of IQOS with HeatStick: Individuals (men and women) between the ages of 40 and 59 (inclusive) with a minimum of 10 pack-year smoking history who switched to and predominantly (>70%) use Heated Tobacco product IQOS/heatstick
  Interventions: Other: Heated Tobacco product IQOS/heatstick
- Smokers of combustible cigarettes: Individuals (men and women) between the ages of 40 and 59 (inclusive) who are currently smoking combustible cigarettes with a minimum of 10 pack-year smoking history
  Interventions: Other: Smoking combustible cigarettes

INTERVENTIONS:
Other: Heated Tobacco product IQOS/heatstick — Heated Tobacco Products: heatsticks heated by iQOS device
  Groups: Users of IQOS with HeatStick
Other: Smoking combustible cigarettes — Current smoking of combustible cigarettes
  Groups: Smokers of combustible cigarettes

SUMMARY:
This study evaluates frequency of exacerbations, respiratory symptoms, physical exercise intolerance and abnormal lung functions among participants who use IQOS with heatsticks compared to smokers of conventional cigarettes

DETAILED DESCRIPTION:
Heated Tobacco Products, such as Heatsticks heated by iQOS device, are specially designed tobacco products that contain tobacco material and several filter sections. Recent studies demonstrate that the vapor from Heatsticks heated by iQOS device contains 90 to 95% less harmful and potentially harmful compounds ("HPHCs") and is 90 to 95% less toxic than the smoke of a reference combustible cigarette.

IQOS with HeatSticks may serve as less risky alternatives to combustible cigarettes and to other traditional tobacco products in clinical setting. The investigators hypothesize that participants using IQOS with HeatSticks will have less prevalent presence of respiratory symptoms, have better functional exercise capacity, and experience less exacerbations compared to those who smoke combustible cigarettes by demonstrating whether the trends of the response variables across time is the same between the exposure and the control groups.

This 5-years observational study includes two cohorts of participants age 40 - 59: (1) smokers of combustible cigarettes (CC smokers -control group) and (2) users of IQOS with HeatStick (exposure group). The study has baseline and periodic (annual) comprehensive clinical assessments, as well as continuous COPD case-finding activities and registering acute exacerbations of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 40-59 years inclusive
* Smoking history ≥10 pack-years (for both cohorts)
* Ability to follow study procedures

Exclusion Criteria:

Pregnant women; Legally incapable individuals;

Patients with history of:

* chronic infectious and non-infectious lung disease except asthma (e.g. pulmonary fibrosis, bronchiectasis, cystic fibrosis, tuberculosis, etc.) diagnosed prior to or during the first visit to KAPM COPD Center;
* previous surgical excision of at least one lung lobe (or having undergone a lung volume reduction procedure);
* active cancer of any localization under treatment;
* suspected cancer of any localization;
* metallic articles in the chest;
* recent eye surgery (during the last 6 month prior to the visit);
* episode (s) of myocardial infarction within less than 6 months prior to the visit or another form of acute or chronic coronary heart disease, history of heart rhythm abnormality with episode of arrhythmia within the last 6 months prior to the visit or long lasting that requires continuous drug therapy;
* acute episode of cerebrovascular ischemic attack within the last 12 month prior to the visit;
* chest or abdominal surgery performed within the last 6 month prior the visit;
* contraindications to salbutamol or refusal to inhale salbutamol;
* chest radiation therapy within the last 12 month prior to the visit; radiology diagnostic procedures of chest within the last 6 months prior to the visit;
* recent (6 weeks before the visit) respiratory tract infection (colds, flus), fever of any etiology with increasing temperature over 37 C at the time of the visit and in the last 2 weeks prior to the visit;
* significant history of alcohol abuse or consumption of more than recommended units of alcohol per week (28 units male and 21 units female);
* positive screening test for HIV antibodies or positive screening for TB, if available at the time of first visit;
* elevated blood pressure (systolic) is ≥160 mmHg at the moment of visit. PMI employees and first degree relatives

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals aged 40 - 59 who live in City of Almaty and smoke combustible cigarettes (CC smokers - control group) or predominantly use IQOS with HeatStick (exposure group).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Presence of respiratory symptoms defined by CAT≥10 | 5 years
  The total COPD Assessment Test Scores 10 and more as an indicator of more symptoms
Functional exercise incapacity | 5 years
  Less than 450 meters walked during the six-minute walk test
Respiratory exacerbations | 5 years
  A worsening of respiratory symptoms, which required treatment with oral corticosteroids or antibiotics, or both or a health care utilization event (office visit, hospital admission, or emergency department visit for a respiratory flare-up).

SECONDARY OUTCOMES:
Evidence of chronic obstructive pulmonary disease | 5 years
  Airflow obstruction based on the fixed ratio of post-bronchodilator FEV1 /FVC < 0.70 criterion
ECG abnormalities | 5 years
  Presence of any ECG abnormalities including pathologic q-waves, ST elevation, ST depression, T-wave inversion, hypertrophy, QRS axis deviation, block, arrhythmia.
Clinical findings by physical pulmonary exam | 5 years
  Presence of any pathological findings during the pulmonary (percussion and inspection) exam
Clinical findings by physical cardiac second sounds exams | 5 years
  Presence of any pathological findings during the cardiac second sounds exam
Metabolic syndrome | 5 years
  Presence of metabolic syndrome based on the IDF definition: Central obesity (defined as waist circumference with ethnicity specific values) PLUS any two of the following four factors: raised triglycerides; reduced HDL cholesterol; raised blood pressure; raised fasting plasma glucose
Decreased Oxygen saturation | 5 years
  Percentage of hemoglobin loaded with oxygen (<95%)
Low Dose Computerised Tomography (LDCT) of the Chest Features | 5 years
  Grading the severity of the following: bronchiectasis, bronchial wall thickening, emphysema, reticular pattern or honeycombing.

CONTACTS AND LOCATIONS:
Overall Officials: Almaz Sharman, MD, PhD, Principal Investigator — Kazakhstan Academy of Preventive Medicine
Locations (1):
- Kazakhstan Academy of Preventive Medicine, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share all participant data except personally identifiable information. Data will be available to open-access after the completion of the study. Access to study data, which is going to be located in our web site, will be granted by request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Sharman A, Zhussupov B, Sharman D, Kim I, Yerenchina E. Lung Function in Users of a Smoke-Free Electronic Device With HeatSticks (iQOS) Versus Smokers of Conventional Cigarettes: Protocol for a Longitudinal Cohort Observational Study. JMIR Res Protoc. 2018 Nov 5;7(11):e10006. doi: 10.2196/10006. PMID 30401669